CLINICAL TRIAL: NCT04464824
Title: Study of the Preventable Passage of Patients Over 75 Years of Age to the Emergency Room of the CHRU of Nancy
Acronym: PE75UN
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Bernadette HANESSE, Principal Investigator, Central Hospital, Nancy, France
Other Study IDs: 2020PI066
Record Dates: First submitted 2020-07-06; First posted 2020-07-09 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Emergencies Elderly

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patient over 75 years of age with an emergency room visit: Patients over 75 years of age, with a visit to the emergency department between April 1, 2019 and September 30, 2019, with a non-hospitalization at the end of their visit to the emergency department.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
The adult emergency service of the Nancy CHRU welcomes an average of 135 visits per day. Approximately 18% are patients over 75 years old, among them 45% go home at the end of their care. The mobile geriatric liaison team intervenes with these patients at the request of the emergency doctors before they return home in order to identify their fragility and implement appropriate measures.

We wish to know the characteristics of these avoidable passages in order to propose preventive measures upstream of these passages. To do this, we need to know the characteristics of those patients with an avoidable passage.

ELIGIBILITY:
Inclusion Criteria:

* age>=75 years old
* admitted at emergency room between first april 2019 and 30 september 2019
* outpatients

Exclusion Criteria:

* inpatients
* discharged patients
* patients discharged against medical advice
* patients brought by police

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: - Patients over 75 years of age, with a visit to the emergency department between April 1, 2019 and September 30, 2019, with a non-hospitalization at the end of their visit to the emergency department.
Sampling Method: Non-Probability Sample
Enrollment: 1573 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-11-23 (Actual); Study Completion 2020-11-23 (Actual)

PRIMARY OUTCOMES:
characteristics of preventable passages to the emergency room of the Nancy CHRU in the population over 75 years old | the day of the admission at emergency room

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Nancy, Nancy, France

IPD SHARING:
Plan to Share IPD: No